CLINICAL TRIAL: NCT06545604
Title: Comprehensive Yoga Therapy Based Lifestyle Prehabilitation Program for Women With Ovarian Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-0374; NCI-2024-06338 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2024-08-05; First posted 2024-08-09 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Yoga; Restraint, Physical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CYT - Prehab Yoga Intervention + ERAS (Experimental)
  Interventions: Other: Yoga Therapy for Nutritional, Physical, and Psychosocial Prehabilitation
- WLC - Wait List Control + ERAS (Experimental)
  Interventions: Other: Usual care supportive services including nutrition counseling per usual care

INTERVENTIONS:
Other: Yoga Therapy for Nutritional, Physical, and Psychosocial Prehabilitation — Two visits per week with a yoga therapist while receiving neoadjuvant chemotherapy to cover dietary counseling, yoga-based movement practices, breathwork practices, mind practices, and behavioral support for the purpose of preparing patients' mind and body for a planned surgery.
  Arms: CYT - Prehab Yoga Intervention + ERAS
Other: Usual care supportive services including nutrition counseling per usual care — Usual care supportive services while receiving neoadjuvant chemotherapy.
  Arms: WLC - Wait List Control + ERAS

SUMMARY:
To provide a comprehensive yoga therapy (CYT) program to patients with ovarian, fallopian tube, or primary peritoneal cancer who are scheduled to receive chemotherapy and then undergo surgery. Researchers want to learn about the effects of the program on patients' quality of life and other outcomes described below.

DETAILED DESCRIPTION:
Primary Objectives:

Primary Objective: to assess the feasibility of a CYT prehabilitation program in women with ovarian cancer scheduled to receive NACT and IDS. Feasibility criteria will include the percent of eligible patients who consent to participate (feasibility is defined as 30% of those approached and are eligible end up consenting) and study retention by the last follow-up (feasibility is defined as 60% of those undergoing surgery remaining in the study and providing some data at baseline and at last follow-up timepoint).

Secondary Objectives:

* Examine the effects of the CYT program on physical conditioning as assessed by the 2-minute step test (2MST) and sit to stand reps (30secSTS) compared with WLC.
* Examine group differences in surgical outcomes including post op stay, readmission rate, post op morbidity, surgical site infection rate, , and time to first chemotherapy post operatively.
* Examine group differences in patient-reported outcomes including QOL, fatigue, stress, sleep disturbances, mental health, social support, and mindfulness.
* Examine if there are group differences in preoperative albumin level, vit D, magnesium levels.
* Examine group differences and changes over time in microbiome biodiversity.
* Examine group differences in body composition (sarcopenia) as measured by routine abdominal CT scans.
* Explore the association between adherence to the components of CYT with ability to sustain behavior changes and between changes in lifestyle parameters with outcomes. This will be explored both within and across groups.

ELIGIBILITY:
Inclusion Criteria:

1. Women with stage III-IV epithelial ovarian, fallopian tube, primary peritonal cancer with recommendations for NACT/IDS at recruitment.
2. Able to read, write, and speak English.
3. 18 years of age or older.
4. Oriented to person, place, and time.
5. Access to internet connection.
6. Access to a tablet, laptop or computer or smart phone.
7. Access and ability to do virtual sessions.

9. Plan for surgical intervention at MD Anderson Cancer Center 9. Performance status 0-2.

Exclusion Criteria:

1. Have completed chemotherapy.
2. Any major thought disorder (e.g., schizophrenia, dementia).
3. Any major communication barriers that would preclude being able to complete the intervention (e.g., visually or hearing impaired).
4. Extreme mobility issues (e.g., unable to get in and out of a chair unassisted).
5. Have a regular mind-body practice or an established yoga practice.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2025-06-06 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
To assess the feasibility of a CYT prehabilitation program in women with ovarian cancer scheduled to receive NACT and IDS. | Through study completion; an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Lois Ramondetta, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org